CLINICAL TRIAL: NCT07189988
Title: Observational Pilot Study to Explore the Social and Health Impacts of a New Model of Care in Oregon: Psilocybin Services on Alcoholism
Status: Active, not recruiting | Type: Observational
Sponsor: Healing Advocacy Fund (Other)
Collaborators: People Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PS13
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder
Keywords: alcoholism; alcohol use disorder
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: All study participants were divided into three cohorts to provide ample time between the participants and facilitators during the psilocybin journey.
  Interventions: Other: psilocybin
- Cohort 2: All study participants were divided into three cohorts to provide ample time between the participants and facilitators during the psilocybin journey.
  Interventions: Other: psilocybin
- Cohort 3: All study participants were divided into three cohorts to provide ample time between the participants and facilitators during the psilocybin journey.
  Interventions: Other: psilocybin

INTERVENTIONS:
Other: psilocybin — All study participants were provided low dose psilocybin.

SUMMARY:
The purpose for this study is to observe the real world experience of participants who are receiving psilocybin in the context of (alcoholism) Alcohol Use Disorder without intervening in the model of care. The study team will engage directly with the participants to examine the outcomes in participants who have been deemed eligible and appropriate to receive psilocybin services at Oregon's Innertrek Patient Service Center (PSC) and who are willing to participate in the People Science pilot study to share their experience concurrently. Since the participant will be making the informed decision to voluntarily take part in this concurrent observational study, there will be no "doctor-patient" relationship between the participant and the People Science Study Investigator.

Study participants will receive the standard of care and medical management from Oregon's Innertrek Patient Service Center facilitators as deemed appropriate per their existing guidelines and practices. People Science will solely be operating as an observer, using an agnostic research data capture system to collect outcomes and follow participant experiences throughout the course of their treatment journey. The study will incorporate participant-reported outcome measures, questionnaires and surveys. The primary endpoint in collecting study data will be to observe the impact of the Psilocybin-Assisted care model on the frequency of heavy drinking days through quantitative and qualitative data analysis for people who struggle with alcohol use. Non-quantitative narratives will also be captured. Throughout the People Science study observations, participants will be in the direct care of the Oregon Patient Service Center facilitators. Findings from this study will contribute knowledge toward the understanding of the use of psilocybin in individuals with self-described alcoholism (AUD).

DETAILED DESCRIPTION:
Alcoholism or Alcohol Use Disorder (AUD) is a chronic and relapsing condition characterized by an inability to control alcohol consumption, leading to significant health, social, and economic consequences. Despite the availability of various treatment modalities, including pharmacotherapies and behavioral interventions, relapse rates remain high, with many individuals failing to achieve long-term abstinence or control. This has spurred interest in exploring novel therapeutic approaches and care models, including the potential use of psychedelic compounds such as psilocybin used in a supportive care environment.

Psilocybin, a naturally occurring psychoactive substance found in certain species of mushrooms, has garnered attention for its potential therapeutic effects in treating mental health disorders such as depression, anxiety, and post-traumatic stress disorder. More recently, research has suggested that psilocybin may be beneficial in addressing substance use disorders, including Alcohol Use Disorder. The mechanism by which psilocybin exerts its effects appears to involve the modulation of neural circuits related to mood regulation, behavior, and self-reflection, which can facilitate profound psychological experiences that may promote lasting changes in behavior and cognition.

Early clinical trials have shown promising results, indicating that psilocybin, when administered in a therapeutic setting, can reduce alcohol consumption and cravings in individuals with Alcohol Use Disorder. In a study published in Journal of American Medical Association of Psychiatry, researchers from New York University Grossman School of Medicine found that heavy alcohol consumption among people with alcohol use disorders was 83 percent lower among participants who had received psilocybin over an 8-month period following the psilocybin administration and almost half of participants who received psilocybin stopped drinking alcohol altogether. These studies highlight the potential for psilocybin to act as a catalyst for psychological insights and behavioral change when combined with psychotherapy or a calming and supportive environment, offering a new avenue for treatment-resistant cases of Alcohol Use Disorder.

In Oregon, excessive alcohol consumption causes 2,000 deaths each year, making it the third leading cause of preventable death in the state. There is a glaring need for support for Oregonians facing alcohol and substance use disorders. Alongside more traditional treatment and harm reduction models, Psilocybin shows promise for treating alcohol and substance disorders. Oregon's state-regulated psilocybin program offers an opportunity to advance real world research on Psilocybin for treating alcohol and substance use disorders.

In 2020, Oregon voters approved a ballot measure (Measure 109) to create the world's first state-regulated psilocybin program to improve the physical, mental, and social well-being of all people. The measure required that the Oregon Health Authority (OHA) create a licensing and regulatory framework for a safe, accessible and equitable program. After a two-year rule making period, licensed service centers are now open and providing psilocybin services to clients in Oregon. Psilocybin services are only delivered in licensed service centers, under the supervision of a trained facilitator, and psilocybin can only be consumed in the service center during that supervised session. There are no retail sales, no off-site consumption, possession, or production of psilocybin (outside of licensed manufacturers).

The sponsor of this pilot research project is the Healing Advocacy Fund (HAF). HAF is a 501c3 non-profit organization that advocates for safe, affordable state-regulated access to psychedelic services. The Healing Advocacy Fund promotes regulations that create a state psilocybin program that is of high quality, accessible, and maximizes safety; educates stakeholders, policymakers, regulators, and the general public on the Oregon psilocybin program; and serves as a convener for the Oregon psilocybin ecosystem to collaboratively address goals and challenges, organize around shared needs, and deliver services to high standards and best practices.

InnerTrek will provide the psilocybin services to individuals who struggle with alcohol use for the pilot. InnerTrek is a psilocybin patient service center located in Portland, Oregon and licensed by the Oregon Health Authority to offer both individual and group psilocybin services, including preparation, administration, and integration sessions.

The position of the People Science research team in this setting is to observe the practices and experiences already occurring in the context of the State of Oregon's Psilocybin Services program at the InnerTrek Patient Service Center. People Science will create the questionnaires to be offered to the participants, as well as analyze data on the observation of participants' perspectives.

ELIGIBILITY:
Inclusion

1. Over 21 years old and reside in Portland, Oregon (all genders)
2. Have a personal smartphone device, internet access, and willing to download Chloe
3. Have been deemed appropriate for care by Oregon's Innertrek Patient Service Center (PSC) and eligible for psilocybin services
4. Willingness to complete study activities and assessments for the duration of the study

Exclusion

Note that #1-3 below are mandatory exclusions for psilocybin-assisted care as directed by the Oregon Health Authority. Any potential participant who:

1. Have a personal history of psychosis per the Oregon Health Authority
2. Have active use of lithium per the Oregon Health Authority
3. Exhibit active thoughts of suicidality per the Oregon Health Authority
4. Are deemed ineligible for psilocybin services by Oregon's Innertrek Patient Service Center (PSC)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited through Oregon's Innertrek Patient Service Center (PSC). They will exhibit struggles with alcoholism or alcohol use disorder, deemed appropriate for care by Oregon's Innertrek Patient Service Center, and eligible for psilocybin services. Once eligibility at the PSC has been determined, eligible participants will be invited to voluntarily participate in the People Science pilot observational research study.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of Heavy Drinking | 12 months
  The primary objective is to study the effects of Oregon Health Authority's (OHA's) psilocybin service program on frequency of heavy drinking among people with alcohol use disorder. This will measured by Percentage of number of heavy drinking days at baseline versus in 30 day increments after completing psilocybin services.

SECONDARY OUTCOMES:
Number of Drinking Days | 12 months
  A secondary objective of this study is to observe the impact of the Oregon Health Authority's Psilocybin program in the context of Alcohol Use Disorder on drinking days. This will be measured by the number of drinking days per month (including heavy and non-heavy drinking).
Days of Complete Abstinence | 12 months
  A secondary objective of this study is to observe the impact of Oregon Health Authority's Psilocybin program in the context of Alcohol Use Disorder on percentage of days of complete abstinence at regular intervals after treatment. This will be measured by the number of days abstinent from alcohol per month.
Diagnostic and Statistical Manual of Mental Disorder (DSM) early remission | 12 months
  A secondary objective of this study is to observe the impact of Oregon Health Authority's Psilocybin program in the context of Alcohol Use Disorder on prevalence of Diagnostic and Statistical Manual of Mental Disorder early remission criteria at regular intervals after treatment. This will be measured by the percentage of participants who meet Diagnostic and Statistical Manual of Mental Disorder early remission criteria at 3 months, and percentage who achieved abstinence at monthly intervals after psilocybin services.
Alcohol Craving | 12 months
  A secondary objective is to observe the impact of Oregon Health Authority's (OHA's) Psilocybin program in the context of Alcohol Use Disorder on subjective alcohol craving. This will be measured by alcohol cravings at the end of each month as measured by the Brief Substance Craving Scale (8-Item).
Spiritual Significance | 12 months
  A secondary objective is to observe the spiritual significance, if any, of participants using Oregon Health Authority's Psilocybin program in the context of Alcohol Use Disorder. This will be measured by the spiritual significance of the program as assessed by the Rating of Spiritual Meaning (FACIT-Sp) questionnaire on a monthly basis.
Treatment Completion Rate | 12 months
  A secondary objective is to evaluate the completion rate of the treatment protocol and any reasons for discontinuation among participants. This will be measured by the percentage of participants who complete the program and reasons for discontinuation on an ongoing basis throughout the course of the 12 month study.
Adverse Events | 12 months
  A secondary objective of the study is to observe the rate of adverse events in Oregon Health Authority's Psilocybin program in the context of Alcohol Use Disorder. This will be measured by the severity and frequency of adverse events assessed weekly during treatment and monthly following treatment.

OTHER OUTCOMES:
Alcohol Abstinence Self-Efficacy | 12 months
  An exploratory objective of the study is to observe the impact of Oregon Health Authority's Psilocybin program in the context of Alcohol Use Disorder on participants' ratings of their own ability to maintain abstinence. This will be measured by the subjective self-efficacy of abstinence as measured by the Alcohol Abstinence Self-Efficacy Scale (AASE) on a monthly basis.
Life Quality | 12 months
  An exploratory objective is to observe the impact of Oregon Health Authority's Psilocybin program in the context of Alcohol Use Disorder on overall quality of life. This will be measured by the Short Form 36 Health Survey, daily optional mood logs, short inventory of problems as well as analysis of participants' notebook entries in Chloe throughout the course of the study and on a monthly basis.
Individual Experiences | 12 months
  An exploratory objective is to assess any individual or cross-cohort themes arising from free text notebook entries by participants. This will be measured by notebook entries in Chloe documenting free-form experiences with and reflections about the intervention throughout the 12 month course of the participant journey.
Alcohol Withdrawal Symptoms | 12 months
  The final exploratory objective of the study is to assess any changes in symptoms of withdrawal from alcohol. This will be measured using a scoring method on the alcohol withdrawal symptom scale weekly and daily basis throughout the 12 month course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft, MD, Principal Investigator — People Science, Inc.
Locations (1):
- Innertrek Patient Service Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will require further internal discussion.